CLINICAL TRIAL: NCT05681806
Title: Assessment of the Efficacy of Carnipure® AAS on Body Composition, Muscle Thickness, and Strength Adaptations in Healthy Men Following a 12-week Strength Training Program
Brief Title: Assessment of the Efficacy of Carnipure® AAS on Body Composition, Muscle Thickness, and Strength Adaptations in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Principal Investigator, Charlie Ottinger, Research Scientist, Applied Science & Performance Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: L091322
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Muscle Hypotrophy
Keywords: Carnipure; Body Composition; Muscle Hypertrophy; Creatine; Muscle Strength
MeSH Terms: conditions — Muscular Atrophy | interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into three parallel groups: two treatment groups of differing Carnipure AAS doses and one active control consuming creatine monohydrate
Masking Description: This is an open label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment High Dose (Experimental): Subjects consuming 1000mg LMP Creatine + 500mg Carnipure crystalline 1x/day
  Interventions: Dietary Supplement: Carnipure AAS
- Treatment Low Dose (Experimental): Subjects consuming 500mg LMP Creatine + 500mg Carnipure crystalline 1x/day
  Interventions: Dietary Supplement: Carnipure AAS
- Active Control (Active Comparator): Subjects consuming 5g creatine monohydrate 1x/day
  Interventions: Dietary Supplement: Creatine Monohydrate

INTERVENTIONS:
Dietary Supplement: Carnipure AAS — A combination of a low dose of Carnipure crystalline (L-carnitine tartrate) and lipid multi-particulate (LMP) creatine monohydrate
  Arms: Treatment High Dose; Treatment Low Dose
Dietary Supplement: Creatine Monohydrate — 5g creatine monohydrate
  Arms: Active Control

SUMMARY:
This study is a 12-week randomized active control trial that is investigating the effects of Carnipure(R) AAS on muscle hypertrophy, body composition, and muscular strength adaptations in healthy men performing a resistance training program.

DETAILED DESCRIPTION:
The study will enroll approximately 45 healthy males (18-40 year old and BMI 18.5-35kg/m2), who are recreationally trained and not presently taking any ergogenic nutritional supplements. Only male subjects will be selected to limit variability in lean mass at baseline as this is the primary variable of interest.

This study will be a 12-week exercise intervention, and will require experienced scientific staff for supervision of subjects. Below are a list of measures to be taken at 0, 6, and 12 weeks.

Primary Measures: these measures will be taken at time 0, 6, and 12-weeks post treatment

* Body composition (Lean and Fat mass) as determined by DXA Secondary Measures: these measures will be taken at time 0, 6, and 12-weeks post treatment
* Pectoral muscle thickness quantification via ultrasonography
* Bench press strength
* Muscle endurance (measured by reps to failure at 50 % 1RM assessed 5 minutes post strength testing)
* Full body strength as assessed by isometric mid thigh pull
* Lower body power as measured by a dual platform ground reaction force plate

Exercise Intervention The exercise intervention will be a 12-week periodized strength training program designed to promote muscle hypertrophy and enhance muscular strength. The 12-weeks will be divided into three 4-week mesocycles in which participants will perform the same exercise routine for 4-weeks before progressing to the next 4-week mesocycle. Participants will train 2x/week with 72-hours of rest between sessions to ensure adequate recovery. All training sessions are designed to last 45-60 minutes (including warmup) and all training sessions will be supervised by a certified personal trainer to ensure proper execution and safety. Two to three minutes of rest will be provided between each set to optimize training adaptations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 18-40 years old
* Recreationally trained (<1-year of training experience)
* Not currently consuming any ergogenic supplements or performance enhancing drugs
* Body mass index (BMI) 18-35 kg/m2
* No recent injuries that would contraindicate participation in a resistance training program
* Willing and able to give written informed consent
* Able to read, understand, sign and date the informed consent document (English only)
* Able and willing to comply with the schedule visit(s) and study requirements.

Exclusion Criteria:

* Currently taking (within the past 30 days) ergogenic dietary supplements including, creatine, protein, amino acids, or stimulants other than caffeine (yohimbe, ephedrine, etc.)
* Currently taking performance enhancing drugs (testosterone or other anabolic-androgenic steroids), human growth hormone, insulin, etc.
* History or current malignancy
* Receiving chemotherapy agents or radiation treatments
* Musculoskeletal disease (muscular dystrophy, arthritis, etc.)
* Recent (<3-months) musculoskeletal injuries
* BMI <18 or >5 kg/m2
* Diagnosis of a terminal illness
* Use of prescription medications that influence muscle anabolism (i.e., prescription hormone therapies, etc.)
* History of alcohol abuse
* History or current drug abuse
* History or current cigarette smoke (including vaping) within the past 14 days from the screening visit
* Insulin-dependent diabetes and/or metformin use
* Chronic kidney or liver disease
* Has significant concurrent illnesses (controlled or uncontrolled), such as diabetes, lupus, epilepsy, or cardiac disorders, hepatitis B/C, HIV, serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years, or other, which in the opinion of the investigator, such conditions might be aggravated as a result of treatment
* The investigator feels that for any reason the subject is not eligible to participate in the study
* History of uncontrolled cardiovascular disease (i.e., myocardial infarction, hypertension, hypercholesterolemia, peripheral vascular disease, other)
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirement and/or record the necessary study measurements
* A family member of the investigator or an employee of the investigator
* Participation in any other investigational study within 30 days prior to consent.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is limited to male participants.
Enrollment: 44 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Body Composition | 12 weeks
  Changes in lean mass and fat mass as measured via dual x-ray absorptiometry

SECONDARY OUTCOMES:
Muscle Hypertrophy | 12 weeks
  Changes in pectoral muscle thickness as measured by b-mode ultrasound
Muscle Strength | 12 weeks
  Changes in bench press 1RM and isometric mid-thigh pull maximum strength
Lower Body Power | 12 weeks
  Changes in lower body power as measured by a dual ground reaction force plate

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Science and Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
All data are owned by the CRO (ASPI) and the sponsor (Lonza Consumer Health).